CLINICAL TRIAL: NCT03380533
Title: The Use of Buprenorphine Transdermal Patches Improves Post-Operative Pain Management in Arthroscopic Rotator Cuff Repair?
Brief Title: Buprenorphine Transdermal Patches in Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, BERNARDO AGUSTIN BERTONA ALTIERI, MD, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2960
Record Dates: First submitted 2017-12-08; First posted 2017-12-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Injury; Analgesics, Opioid; Buprenorphine
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Buprenorphine; Tramadol

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine Patch (Active Comparator): Buprenorphine 10mg Patch + Placebo Tablet + Multimodal Oral Scheme
  Multimodal Oral Scheme:
  Diclofenac 75mg c 12h Rescues with tramadol 50 mg (maximum rescue dose 150mg, minimum frequency between rescues 4hs)
  Interventions: Drug: Buprenorphine; Drug: Multimodal Oral Scheme; Drug: Placebo Tablet
- Tramadol Tablet (Active Comparator): Placebo Patch + Tramadol 50mg Tablet + Multimodal Oral Scheme
  Multimodal Oral Scheme:
  Diclofenac 75mg c 12h Rescues with tramadol 50 mg (maximum rescue dose 150mg, minimum frequency between rescues 4hs)
  Interventions: Drug: Placebo Patch; Drug: Multimodal Oral Scheme; Drug: Tramadol

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine 10mg transdermal patch used during the first five postoperative days after arthroscopic rotator cuff repair
  Other Names: Buprenorphine Patch
  Arms: Buprenorphine Patch
Drug: Placebo Patch — Adhesive patch with the same macroscopic characteristics to the buprenorphine patch, without drugs.
  Arms: Tramadol Tablet
Drug: Multimodal Oral Scheme — Diclofenac 75mg c 12h Tramadol 50mg c 12h. Rescues with tramadol 50 mg (maximum rescue dose 150mg, minimum frequency between rescues 4hs)
Drug: Tramadol — Tramadol 50mg tablet that the patient consumes every 8 hours during the first five days
  Other Names: Tramadol Tablet
  Arms: Tramadol Tablet
Drug: Placebo Tablet — Placebo tablet that the patient consumes every 8 hours during the first five days
  Arms: Buprenorphine Patch

SUMMARY:
Arthroscopic rotator cuff repair is associated with poor post-operative pain management. The multimodal analgesic scheme (oral non-steroidal anti-inflammatory drugs associated with oral opioids) currently used according to the pain management guidelines is insufficient for most of these patients.

There are few reports on the use of buprenorphine in post-operative pain with encouraging results. There is no evidence of its use in the management of post-operative pain of arthroscopic rotator cuff repair

DETAILED DESCRIPTION:
Traditionally, oral opioids have been used to manage the postoperative pain of arthroscopic rotator cuff repair (ARCR) . Due to the intensity of pain, it often requires high doses of opioids, frequently associated with side effects, such as nausea, vomiting, constipation, disorientation, among others, which, in the context of an outpatient, interfere with the postoperative period, sometimes resulting in hospital readmissions. due to both the poor management of pain and the adverse effects of opioids.

Although there are invasive strategies of analgesia, such as the placement of continuous infusion catheters of analgesics in the sub-acromial space, these are methods that demand the management of the devices, in some cases requiring prolongation of hospitalization for the patient. management of the same, without being exempt from complications as any analgesic method added to those related to the method.

Currently, the post-operative analgesia strategy widely accepted globally and that used in our center, is multimodal analgesia, in which NSAIDs (Anti-Inflammatory Non-Steroids) and oral opioids are associated. A combination of both analgesic mechanisms of action is used as a basic scheme, and rescues with opioids are carried out orally. Although the literature supports its cost-benefit, this approach is often insufficient, not achieving adequate control of postoperative pain in ARCR, with 64% of our patients reporting poor pain management in the first week of post-operative and 10% that require re-entry to day hospital for pain management.

The application of transdermal opioid release patches is a method of non-invasive analgesia, which has previously been used with good results for the management of postoperative pain. In ARCR there is no evidence of its use in the management of post-operative pain The main advantages could be related to the plasma stability of the drug (buprenorphine), which implies fewer peaks and valleys of analgesia, a better compliance by the patient since it is of weekly duration and lower incidence of cognitive deterioration related to other opioids.

Compared with other opioids, buprenorphine is associated with a lower risk of abuse, overdose and poisoning due to the ceiling effect. Despite this favorable pharmacological profile, the use of buprenorphine in patches has a lower abuse rate than other forms of administering the same drug. On the one hand, the release rate of the patch may be insufficient to satisfy the compulsive desire and, to that end, the patch may be less desirable. On the other hand, the availability in the market and the way to use the patches could be other conditioning factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with rotator cuff injury, regardless of the type of injury.
* Patient undergoing Arthroscopic Rotator Cuff Repair

Exclusion Criteria:

1. Refusal to participate or inability to understand the informed consent process.
2. Inability to understand subjective scales of pain
3. Regular use of narcotics
4. Allergy or intolerance to drugs used in the protocol
5. Consumption of drugs that interact with Buprenorphine (anticholinergics, Atropine, Belladonna, Benztropine, Dicyclomine, Diphenhydramine, Isopropamide, Procyclidine and Scopolamine, Antiarrhythmics, Amiodarone, Disopyramide, Dofetilide, Procainamide, Quinidine and Sotalol.

   Anticonvulsants; Carbamazepine, Phenobarbital, Phenytoin and Rifampin)
6. History of previous surgeries in shoulder treated with RAMR
7. Previous neuromuscular deficit
8. Febrile Syndrome
9. Autoimmune or Rheumatologic Disease
10. History of intestinal transit disorders (paralytic ileus)
11. History of alcohol or drug abuse
12. Patients in psychological or psychiatric treatment for anxiety disorders, personality disorders, mood disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Pain perception | Five days
  subjective perception of pain through the use of an analogous visual scale

SECONDARY OUTCOMES:
Consumption of rescue opiods | Five Days
  consumption of rescue opiods
Hours of sleep | 5 days
  hours of sleep
Perception of Sickness | 5 days
  presence or not of nausea
Readmissions rate | 5 days
  record of hospital readmissions for pain or complications related to the use of buprenorphine patches
Misuse or abuse of opioids rate | Fourth month post operatory
  Behaviors of misuse or abuse of opioids after the immediate postoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided